CLINICAL TRIAL: NCT01553344
Title: Serum Sclerostin Level in Patients With Vitamin D Deficiency
Brief Title: Serum Sclerostin Level & Treatment of Vitamin D Deficiency
Acronym: OMSOST
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan Karacan, Clinical Associated Professor, Chief of Physical Med & Rehab Clinic, Bagcilar Training and Research Hospital
Other Study IDs: BEAH FTR -7
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Endocrine System Diseases; Vitamin D Deficiency
Keywords: sclerostin; osteomalacia; vitamin D deficiency
MeSH Terms: conditions — Endocrine System Diseases; Vitamin D Deficiency; Sclerosteosis; Osteomalacia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to determine serum sclerostin levels and change in serum sclerostin levels in patients with Vitamin D deficiency treated with calcium and vitamin D.

Healthy premenopausal Patients with Vitamin D deficiency diagnosed and routinely treated with calcium and vitamin D will be included in the study. This is an observational study. The serum sclerostin levels will be measured before and after Vitamin D treatment.

DETAILED DESCRIPTION:
This study is a prospective, observational, single-center study. Ethical approval was obtained from the Institutional Review Board.

This study will be completed with patients with Vitamin D deficiency. An intravenous cannula will be inserted into the antecubital vein. Blood samples will be obtained before and after treatment.

Serum will be collected and will be centrifuged for 15 minutes at 1000Xg within 30 minutes of collection. Aliquots of serum will be added to eppendorf tubes and stored at -20°C.

Serum sclerostin levels will be measured using a Human Sclerostin ELISA kit (Cusabio, Catalog No: CSB-E13146h, Newark, DE, USA). All assays will be performed according to the manufacturer's instructions. The minimum detectable concentration of human sclerostin is typically <0.012 ng/ml. Intra-assay precision is less than 8%.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Serum 25(OH)D < 10 ng/mL

Exclusion Criteria:

* Anemia
* Tumor-induced osteomalacia (hypophosphatemia)
* Hypothyroidism
* Hepatic / renal disease
* Primary hyperparathyroidism
* Fibromyalgia
* Polymyalgia rheumatica
* Serum 25(OH)D > 10 ng/mL
* Vitamin D and calcium treatment commenced prior to study participation

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with vitamin D deficiency
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Serum sclerostin level | 8 weeks
  Changes in serum sclerostin level in patients with osteomalacia who are scheduled for routine treatment of osteomalacia

CONTACTS AND LOCATIONS:
Overall Officials: MUHARREM CIDEM, MD, Principal Investigator — Bagcilar Training & Research Hospital Istanbul, Turkey
Locations (1):
- Bagcilar Training & Research Hospital, Istanbul, Turkey (Türkiye)